CLINICAL TRIAL: NCT04740281
Title: Footwear Among Medical Doctors: An Observational Study of Fashion in Footwear Between Subspecialties
Brief Title: Footwear Among Medical Doctors
Acronym: TÅFIS
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CLOGS21
Record Dates: First submitted 2021-02-01; First posted 2021-02-05 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-01

CONDITIONS: Shoes
Keywords: Footwear; Fashion; Medical doctors; Clogs
MeSH Terms: interventions — Shoes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Medical Doctors at Aarhus University Hospital, Denmark: Medical Doctors from different subspecialties at Aarhus University Hospital, Denmark. Blinded for the purpose of the trial, their footwear will be evaluated by trial responsible personal.
  Interventions: Behavioral: Footwear

INTERVENTIONS:
Behavioral: Footwear — Assessment of footwear
  Other Names: Shoes

SUMMARY:
The footwear fashion among medical doctors has been static for decades with a high preference for clogs. However, other types of shoes have been introduced, including sneakers, sandals etc. In some subspecialties with a "need-for-speed", high-agility footwear may be prioritized, while other subspecialist may benefit from "easy-to-clean" shoes. Even comfortability may influence the choice of footwear.

We intend to investigate measures of footwear fashion among medical doctors working at Aarhus University Hospital, Denmark. Participants will be blinded.

ELIGIBILITY:
Inclusion Criteria:

* Medical Doctor working at Aarhus University Hospital, Denmark
* Wear shoes at work
* Presence at the randomly selected meetings for medical doctors, where trial personal will perform the footwear assessment.

Exclusion Criteria:

* Medical student
* Nurse or other health care profession
* Unidentifiable gender and/or educational level

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Medical Doctors working at Aarhus University Hospital, Denmark. The participants will be divided into two groups: Doctors in specialization (In Danish; KBU-, Intro- and HU-læger) and senior doctors (Specialists).
Sampling Method: Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Footwear preference by subspecialty | Assessed in the data collection period - Spring 2021
  Differences in footwear between medical subspecialties

SECONDARY OUTCOMES:
Footwear preference by seniority | Assessed in the data collection period - Spring 2021
  Differences in footwear of medical doctors by seniority
Footwear preference by sex | Assessed in the data collection period - Spring 2021
  Differences in footwear between male and female doctors

CONTACTS AND LOCATIONS:
Overall Officials: Rasmus H Gantzel, MD, Principal Investigator — Department of Hepatology and Gastroenterology, Aarhus University Hospital; Mikkel B Kjær, Study Director — Department of Hepatology and Gastroenterology, Aarhus University Hospital; Kristoffer Kjærgaard, Study Chair — Department of Hepatology and Gastroenterology, Aarhus University Hospital
Locations (1):
- Department of Hepatology and Gastroenterology, Aarhus University Hospital, Aarhus N, Central Jutland, Denmark

REFERENCES:
- [Derived] Gantzel RH, Kjaer MB, Kjaergaard K. [Christmas article: Footwear fashion amongst medical doctors - are clogs fashion or history?]. Ugeskr Laeger. 2021 Dec 13;183(50):V20214. Danish. PMID 34895430